CLINICAL TRIAL: NCT02034578
Title: Study of Apixaban Oral Solution Bioavailability When Administered Through a Nasogastric Tube in Healthy Subjects
Brief Title: Phase 1 Oral Solution Bioavailability Study of Apixaban When Administered Through a Nasogastric Tube in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CV185-091
Record Dates: First submitted 2014-01-10; First posted 2014-01-13 (Estimated); Results first posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A: Apixaban (Experimental): Single dose Apixaban 5 mg (0.4 mg/mL x 12.5 mL) oral solution via oral syringe
  Interventions: Drug: Apixaban
- Arm B: Apixaban (Experimental): Single dose Apixaban 5 mg (0.4 mg/mL x 12.5 mL) oral solution via nasogastric tube (NGT) immediately followed by 60 mL of D5W via NGT
  Interventions: Drug: Apixaban
- Arm C: Apixaban (Experimental): Single dose Apixaban 5 mg (0.4 mg/mL x 12.5 mL) oral solution via NGT immediately followed by 60 mL of infant formula via NGT
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban
  Other Names: BMS-562247

SUMMARY:
The purpose of this study is to assess the bioavailability of Apixaban solution administered through NGT and washed with Dextrose 5% in water (D5W) or infant formula relative to Apixaban solution administered orally in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

- Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Any history or evidence of abnormal bleeding or coagulation disorders, intracranial hemorrhage, or abnormal bleeding (including heavy menstrual bleeding that has resulted in anemia within the past 1 year) or coagulation disorders in a first degree relative

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Parexel Baltimore Early Phase Clinical Unit, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Song Y, Wang X, Perlstein I, Wang J, Badawy S, Frost C, LaCreta F. Relative Bioavailability of Apixaban Solution or Crushed Tablet Formulations Administered by Mouth or Nasogastric Tube in Healthy Subjects. Clin Ther. 2015 Aug;37(8):1703-12. doi: 10.1016/j.clinthera.2015.05.497. Epub 2015 Jul 15. PMID 26188837
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were admitted to the clinical facility on the evening prior to dosing (Day -1) and remained confined to the clinic for the duration of study.
Pre-assignment Details: 75 enrolled; 21 randomized; 21 treated. Of the 54 not treated: 47 no longer met study criteria, 1 not needed due to adequate number of participants, 3 withdrew consent, 1 died due to substance abuse, 1 no show, 1 discharged as alternate. Study was 3-treatment crossover administered over 3 periods. ≥4 days washout after doses in Periods 1 and 2.
Groups:
- Treatment A, Then Treatment B, Then Treatment C; Treatment A, Then Treatment C, Then Treatment B; Treatment B, Then Treatment A, Then Treatment C; Treatment B, Then Treatment C, Then Treatment A; Treatment C, Then Treatment A, Then Treatment B; Treatment C, Then Treatment B, Then Treatment A: Treatment A: Single dose apixaban 5 mg (0.4 mg/mL oral solution x 12.5 mL) administered by mouth via oral syringe.
  Treatment B: Single dose apixaban 5 mg (0.4 mg/mL oral solution x 12.5 mL) administered via a Nasogastric tube (NGT) immediately followed by 60 mL of dextrose 5% in water (D5W) via NGT.
  Treatment C: Single dose apixaban 5 mg (0.4 mg/mL oral solution x 12.5 mL) administered via an NGT immediately followed by 60 mL of infant formula via NGT.
  After a 10 hour fast, on Day 1 of Period 1, participants were randomized to one of six treatment sequences across 3 periods(ABC, ACB, BAC, BCA, CAB or CBA). Fasted participants received a single dose of apixaban 5 mg on Day 1 of Periods 1, 2, and 3. After participants received the Period 1 dose, there was ≥4-days of washout before their Period 2, Day 1 dose was administered, which was followed by another ≥4-days of washout. After their Period 3, Day 1 dose, participants were discharged on Day 4 of Period 3.
Period: Overall Study
Arm/Group | Treatment A, Then Treatment B, Then Treatment C | Treatment A, Then Treatment C, Then Treatment B | Treatment B, Then Treatment A, Then Treatment C | Treatment B, Then Treatment C, Then Treatment A | Treatment C, Then Treatment A, Then Treatment B | Treatment C, Then Treatment B, Then Treatment A
Started | 4 | 3 | 4 | 3 | 4 | 3
Completed | 4 | 3 | 4 | 3 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received study drug were analyzed.
Groups:
- 5mg Apixaban: After a 10 hour fast, participants were randomized to one of six treatment sequences (ABC, ACB, BAC, BCA, CAB or CBA) administered over 3 periods. Fasted participants received a single dose of apixaban 5 mg on Day 1 of Periods 1, 2, and 3. Treatment A was administered via oral syringe, Treatment B was administered via an NGT followed by 60 mL of D5W via an NGT, and Treatment C was administered via an NGT, followed by 60 mL of infant formula via an NGT. There was at least a 4 day washout before receiving the next scheduled treatment in the next period.
Arm/Group | 5mg Apixaban
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Discontinuation Due to AEs, Death
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: Day 1 to Day 12
Population: All participants who received study drug were analyzed.
Measure: Number; unit: participants
Groups:
- 5mg Apixaban Via Oral Syringe (A): Single dose Apixaban 5 mg oral solution via oral syringe
- 5mg Apixaban Via NGT Followed by D5W (B): Single dose Apixaban 5 mg oral solution via NGT immediately followed by 60 mL of D5W via NGT
- 5 mg Apixaban Via NGT Followed by Infant Formula (C): Single dose Apixaban 5 mg oral solution via NGT immediately followed by 60 mL of infant formula via NGT
Arm/Group | 5mg Apixaban Via Oral Syringe (A) | 5mg Apixaban Via NGT Followed by D5W (B) | 5 mg Apixaban Via NGT Followed by Infant Formula (C)
Number analyzed (Participants) | 21 | 21 | 21
participants
  Discontinuation Due to AE | 0 | 0 | 0
  SAE | 0 | 0 | 0
  Death | 0 | 0 | 0
  Adverse Events | 2 | 4 | 3

2. Primary Outcome: Adjusted Geometric Mean Maximum Observed Plasma Concentration (Cmax) of Apixaban
Description: Samples of plasma from participants were obtained at the following times: 0 hour (h) and post dose at 0.25h, 0.50h, 1h, 2h, 3h, 4h, 5h, 6h, 9h, 12h, 24h, 36h, 48h, 60h, and 72h. Apixaban was assayed using a validated Liquid chromatography tandem mass spectrometry (LC-MS/MS) method during the period of known analyte stability. Maximum observed plasma concentration (Cmax) was measured in nanograms per milliliter (ng/mL).
Time Frame: Day 1 (0 h, 0.25h, 0.50h, 1h, 2h, 3h, 4h, 5h, 6h, 9h, 12h, 24h, 36h, 48h, 60h, and 72h post dose) in Periods 1, 2 and 3
Population: All participants who received study drug and had adequate PK profiles were included in the analysis.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | 5mg Apixaban Via Oral Syringe (A) | 5mg Apixaban Via NGT Followed by D5W (B) | 5 mg Apixaban Via NGT Followed by Infant Formula (C)
Number analyzed (Participants) | 21 | 21 | 21
ng/mL | 190.873 [176.032 to 206.965] | 181.862 [162.834 to 203.112] | 153.693 [140.686 to 167.904]
Statistical Analysis 1: Comparison: 5mg Apixaban Via Oral Syringe (A) vs 5mg Apixaban Via NGT Followed by D5W (B); B versus A; Test type: Superiority or Other; Ratio of adjusted geometric means = 0.953, 90% CI 2-sided [0.873 to 1.040]
Statistical Analysis 2: Comparison: 5mg Apixaban Via Oral Syringe (A) vs 5 mg Apixaban Via NGT Followed by Infant Formula (C); C versus A; Test type: Superiority or Other; Ratio of adjusted geometric means = 0.805, 90% CI 2-sided [0.749 to 0.865]

3. Secondary Outcome: Median Time of Maximum Observed Plasma Concentration (Tmax) of Apixaban
Description: Samples of plasma from participants were obtained at the following times: 0 hour (h), 0.25h, 0.50h, 1h, 2h, 3h, 4h, 5h, 6h, 9h, 12h, 24h, 36h, 48h, 60h, and 72h, relative to the single dose on Day 1 in each cross over period. Apixaban was assayed using a validated LC-MS/MS method during the period of known analyte stability. Maximum observed plasma concentration (Tmax) was measured in hours (h).
Time Frame: Day 1 (0 h, 0.25h, 0.50h, 1h, 2h, 3h, 4h, 5h, 6h, 9h, 12h, 24h, 36h, 48h, 60h, and 72h post dose) in Periods 1, 2 and 3
Measure: Median (Full Range); unit: h
Arm/Group | 5mg Apixaban Via Oral Syringe (A) | 5mg Apixaban Via NGT Followed by D5W (B) | 5 mg Apixaban Via NGT Followed by Infant Formula (C)
Number analyzed (Participants) | 21 | 21 | 21
h | 0.517 [0.48 to 2.00] | 1.000 [0.30 to 2.00] | 1.00 [0.48 to 2.00]

4. Secondary Outcome: Adjusted Geometric Mean Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of Last Quantifiable Plasma Concentration, AUC(0-T), of Apixaban
Description: Samples of plasma from participants were obtained at the following times: 0 h, 0.25h, 0.50h, 1h, 2h, 3h, 4h, 5h, 6h, 9h, 12h, 24h, 36h, 48h, 60h, and 72h, relative to the single dose on Day 1 in each cross over period. Apixaban was assayed using a validated LC-MS/MS method during the period of known analyte stability. AUC(0-T) was measured in nanograms*hours per milliliter (ng*h/mL).
Time Frame: Day 1 (0 h, 0.25h, 0.50h, 1h, 2h, 3h, 4h, 5h, 6h, 9h, 12h, 24h, 36h, 48h, 60h, and 72h post dose) in Periods 1, 2 and 3
Population: All participants who received study drug and had adequate PK profiles were included in the analysis.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | 5mg Apixaban Via Oral Syringe (A) | 5mg Apixaban Via NGT Followed by D5W (B) | 5 mg Apixaban Via NGT Followed by Infant Formula (C)
Number analyzed (Participants) | 21 | 21 | 21
ng*h/mL | 1269.784 [1140.000 to 1414.343] | 1226.339 [1064.999 to 1412.121] | 1166.572 [1031.549 to 1319.268]
Statistical Analysis 1: Comparison: 5mg Apixaban Via Oral Syringe (A) vs 5mg Apixaban Via NGT Followed by D5W (B); B versus A; Test type: Superiority or Other; Ratio of adjusted geometric means = 0.966, 90% CI 2-sided [0.924 to 1.010]
Statistical Analysis 2: Comparison: 5mg Apixaban Via Oral Syringe (A) vs 5 mg Apixaban Via NGT Followed by Infant Formula (C); C versus A; Test type: Superiority or Other; Ratio of adjusted geometric means = 0.919, 90% CI 2-sided [0.896 to 0.942]

5. Secondary Outcome: Adjusted Geometric Mean Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time, AUC(INF), of Apixaban
Description: Samples of plasma from participants were obtained at the following times: 0 h, 0.25h, 0.50h, 1h, 2h, 3h, 4h, 5h, 6h, 9h, 12h, 24h, 36h, 48h, 60h, and 72h, relative to the single dose on Day 1 in each cross over period. Apixaban was assayed using a validated LC-MS/MS method during the period of known analyte stability. AUC(0-INF) was measured in ng*h/mL.
Time Frame: Day 1 (0 h, 0.25h, 0.50h, 1h, 2h, 3h, 4h, 5h, 6h, 9h, 12h, 24h, 36h, 48h, 60h, and 72h post dose) in Periods 1, 2 and 3
Population: All participants who received study drug and had adequate PK profiles were included in the analysis.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | 5mg Apixaban Via Oral Syringe (A) | 5mg Apixaban Via NGT Followed by D5W (B) | 5 mg Apixaban Via NGT Followed by Infant Formula (C)
Number analyzed (Participants) | 21 | 21 | 21
ng*h/mL | 1292.775 [1161.691 to 1438.650] | 1250.913 [1088.380 to 1437.718] | 1192.387 [1056.600 to 1345.624]
Statistical Analysis 1: Comparison: 5mg Apixaban Via Oral Syringe (A) vs 5mg Apixaban Via NGT Followed by D5W (B); B versus A; Test type: Superiority or Other; Ratio of adjusted geometric means = 0.968, 90% CI 2-sided [0.926 to 1.011]
Statistical Analysis 2: Comparison: 5mg Apixaban Via Oral Syringe (A) vs 5 mg Apixaban Via NGT Followed by Infant Formula (C); C versus A; Test type: Superiority or Other; Ratio of adjusted geometric means = 0.922, 90% CI 2-sided [0.899 to 0.947]

6. Secondary Outcome: Mean Plasma Elimination Half-Life (T-HALF) of Apixaban
Description: Samples of plasma from participants were obtained at the following times: 0 h, 0.25h, 0.50h, 1h, 2h, 3h, 4h, 5h, 6h, 9h, 12h, 24h, 36h, 48h, 60h, and 72h, relative to the single dose on Day 1 in each cross over period. Apixaban was assayed using a validated LC-MS/MS method during the period of known analyte stability. T-HALF was measured in hours (h).
Time Frame: Day 1 (0 h, 0.25h, 0.50h, 1h, 2h, 3h, 4h, 5h, 6h, 9h, 12h, 24h, 36h, 48h, 60h, and 72h post dose) in Periods 1, 2 and 3
Population: All participants who received study drug and had adequate PK profiles were included in the analysis.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 5mg Apixaban Via Oral Syringe (A) | 5mg Apixaban Via NGT Followed by D5W (B) | 5 mg Apixaban Via NGT Followed by Infant Formula (C)
Number analyzed (Participants) | 21 | 21 | 21
h | 10.5 (4.2) | 10.4 (4.5) | 10.6 (3.8)

7. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram, Vital Sign, or Physical Examination Findings
Description: 12-lead electrocardiograms (ECGs) and Vital Signs were performed at Screening, and Day 1 of Periods 1, 2 and 3 (pre-dose and prior to NGT placement, if done). Vital signs and ECGs were also performed on Day 4 of Period 3, prior to discharge from the study. Vital signs included body temperature, respiratory rate, seated blood pressure and heart rate. Blood pressure and heart rate were measured after the participant had been seated quietly for at least 5 minutes. Participants had physical examinations on Period 1, Day 1 (pre-dose) and Day 4 of Period 3, prior to study discharge.
Time Frame: Screening, Day 1 of Periods, 1, 2, and 3, and Day 4 of Period 3
Population: All participants who received study drug were analyzed.
Measure: Number; unit: participants
Arm/Group | 5mg Apixaban Via Oral Syringe (A) | 5mg Apixaban Via NGT Followed by D5W (B) | 5 mg Apixaban Via NGT Followed by Infant Formula (C)
Number analyzed (Participants) | 21 | 21 | 21
participants
  ECG | 0 | 0 | 0
  Vital Signs | 0 | 0 | 0
  Physical Examination | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Marked Abnormality in Hematology, Chemistry and Urinalysis Laboratory Tests
Description: Participants were required to fast for at least 10 hours prior to the collection of specimens for clinical laboratory tests. Tests were performed at Screening, Day -1, and Day 4 of each period 1 - 3. Leukocyte criteria: Lower limits of normal (LLN), upper limits of normal (ULN), pre-treatment (preRX). Low Leukocytes: if value < 0.9*LLN, or if preRX < LLN then use < 0.85* preRX. High lymphocytes: if value > 7.500 10^3 cells/ µL. Low neutrophils plus bands: if value <= 1.500 10^3 cells/µL. High creatine kinase: if value > 1.5* ULN. Blood in urine: if value >= 2 plus, or if preRX >= 1 plus then use >= 2*preRX.
Time Frame: Screening, Day -1, Day 4 of Periods, 1, 2, and 3
Population: Participants who received study drug were analyzed.
Measure: Number; unit: participants
Groups:
- 5mg Apixaban: After a 10 hour fast, participants were randomized on Day 1 of Period 1 to one of six treatment sequences (ABC, ACB, BAC, BCA, CAB or CBA) and received a single dose of apixaban 5 mg. Treatment A was administered via oral syringe, Treatment B was administered via an NGT followed by 60 mL of D5W via an NGT, and Treatment C was administered via an NGT, followed by 60 mL of infant formula via an NGT. There was at least a 4 day washout before receiving the next scheduled treatment in Period 2 and Period 3.
Arm/Group | 5mg Apixaban
Number analyzed (Participants) | 21
participants
  Low Leukocytes | 1
  High Lymphocytes | 1
  Low Neutrophils plus bands | 5
  High Creatine Kinase | 1
  Blood in Urine | 1

ADVERSE EVENTS:
Time Frame: Day 1 to Day 12
Description: All participants who received at least one dose of study drug were analyzed.
Groups:
- 5mg Apixaban Via Oral Syringe (A): After a 10 hour fast, on Day 1 of Period 1, participants were randomized to one of six treatment sequences administered over 3 Periods (ABC, ACB, BAC, BCA, CAB or CBA) and received a single dose of apixaban 5 mg. After participants received the Period 1 dose, there was ≥4-days of washout before their Period 2, Day 1 dose was administered, which was followed by another ≥4-days of washout. After their Period 3, Day 1 dose, participants were discharged on Day 4 of Period 3.
  In Treatment A the single dose of 5 mg apixaban was administered via oral syringe.
- 5mg Apixaban Via NGT Followed by D5W (B): In Treatment B the single dose of 5 mg apixaban was administered via nasogastric tube (NGT) followed by 60 mL of dextrose, water (D5W) via the NGT.
- 5 mg Apixaban Via NGT Followed by Infant Formula (C): In Treatment C, the single dose of 5 mg apixaban was administered via NGT, followed by 60 mL of infant formula via the NGT.
Arm/Group | 5mg Apixaban Via Oral Syringe (A) | 5mg Apixaban Via NGT Followed by D5W (B) | 5 mg Apixaban Via NGT Followed by Infant Formula (C)
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 2/21 | 4/21 | 3/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5mg Apixaban Via Oral Syringe (A) (N=21) | 5mg Apixaban Via NGT Followed by D5W (B) (N=21) | 5 mg Apixaban Via NGT Followed by Infant Formula (C) (N=21)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 0
Eyelid Oedema (Eye disorders) | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trials primary publication.